CLINICAL TRIAL: NCT05064917
Title: Basophil Activation Test (BAT) Cow's Milk as a Replacement for the Expensive, Burdensome and Risky Food Challenge Tes
Brief Title: BAT Cow's Milk for the Replacement of the Food Challenge Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: Alrijne Hospital (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Bernhoven Hospital (Other); Catharina Ziekenhuis Eindhoven (Other); Elkerliek Hospital (Other); Erasmus Medical Center (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Maasstadziekenhuis (Unknown); Meander Medisch Centrum (Other); OLVG (Network); Spaarne Gasthuis (Other); Franciscus Gasthuis (Other); University Medical Center Groningen (Other); UMC Utrecht (Other); Viecurie Medisch Centrum voor Noord LImburg (Unknown); Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: NL76893.091.21
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Cow Milk Allergy
Keywords: Basophil Activation test; Cow's milk; oral food challenge
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with suspected cow's milk allergy
  Interventions: Diagnostic Test: Blood draw

INTERVENTIONS:
Diagnostic Test: Blood draw — The burden for child/parents in this study is low as it is limited to a single blood draw, which is already necessary for usual diagnostic care in about 70% of the children

SUMMARY:
The prevalence of children suspected of a cow's milk allergy is 17% in the Netherlands. Cow's milk diagnosis is based on a food challenge test However, this food challenge test is expensive, time consuming, risky, with waiting lists of several months. This waiting time results in unnecessarily long-term use of expensive hypoallergenic milk formula Therefore, there is a great need to introduce a better and faster diagnostic test for cow's milk allergy diagnosis in standard care. The in vitro Basophil Activation Test (BAT) is cheap, quick (result < 1 day, no waiting list), safe for the child and is a reliable alternative for the food challenge test to diagnose an IgE-mediated allergy. A diagnostic work-up with the BAT is expected to achieve a relevant reduction in the number of expensive and risky food challenges and the prescription of hypoallergenic formula. The reduction in diagnostic delay will increase quality of life.

Objective: Determination of the (cost)effectiveness of the replacement of the expensive, risky and time-consuming food challenge test by the Basophil Activation Test (BAT) for the diagnosis of an IgE-mediated cow's milk allergy in children.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-12 years
2. Suspected of cow's milk allergy with one or more of the following complaints after intake of cow's milk:

   * angioedema
   * urticaria
   * sneezing and rhinitis <2 hours after feeding
   * sensation of swelling in the throat and/or difficulty swallowing <2 hours after feeding
   * voice change/hoarseness <2 hours after feeding
   * cough <2 hours after feeding
   * wheezing and/or shortness of breath <2 hours after feeding
   * loss of consciousness <2 hours after feeding
   * vomiting or abdominal pain or diarrhoea <2 hours after feeding in children <4 years only in combination with IgE-mediated complaints in other tracts
3. Placed on a waiting list for a hospital food challenge test
4. Blood draw for cow's milk sIgE and BAT < 3 months before the food challenge test. This blood draw will be simultaneously scheduled with a blood draw for regular diagnostics.
5. Signed informed consent parents/guardians

Exclusion Criteria:

1. Age > 12 years
2. Suspicion of Food Protein-Induced Enterocolitis Syndrome (FPIES)
3. Eosinophilic esophagitis due to a cow's milk allergy
4. Suspected cow's milk allergy <4 years with crying and/or agitation and/or eczema and/or abdominal pain and/or failure to thrive and/or blood loss per anum and/or diarrhoea and/or reflux and/or vomiting as the only manifestation of the allergy without IgE-mediated symptoms in another organ system
5. Systemic immunosuppressant use
6. Other underlying chronic conditions (immunological, oncological, chromosomal abnormalities).

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children suspected of an IgE-mediated cow's milk allergy and are eligible for a food challenge test at 2nd and 3rd line allergy centres.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the in vitro Basophil Activation Test (BAT) Cow's Milk | 3 months

SECONDARY OUTCOMES:
Cost-effectiveness of the BAT cow's milk | 1 year
  Cost-effectiveness of the BAT cow's milk compared to the food challenge test
Food allergy Quality of life | Before and one month after the food challenge test
  Quality of life measured by The Food Allergy Quality of Life Questionnaire (FAQLQ-CF)
Health related Quality of life | Before and one month after the food challenge test
  Quality of life measured by Kidscreen-10

CONTACTS AND LOCATIONS:
Locations (1):
- Janneke Ruinemans, Arnhem, Gelderland, Netherlands